CLINICAL TRIAL: NCT00296751
Title: Epidural Analgesia Versus IV Meperidine for Labor Pain Control. Objective Evaluation of the Pain Intensity Influence on the Autonomic Nervous System.
Brief Title: Epidural Analgesia Versus IV Meperidine for Labor Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: epiduralCTIL
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2008-04

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Fentanyl

INTERVENTIONS:
Procedure: ECG recording
Procedure: Epidural catheter insertion
Drug: Intravenous meperidine injection
Drug: Epidural Bupivacaine and fentanyl injection

SUMMARY:
60 female that care for pain control during second stage of delivery, will choose between epidural or systemic analgesia. Continuous ECG (3 lead)monitoring will be recorded during the second stage for 10 minutes. 30 minutes after administration of either pain relief, a second recording of maternal ECG will take place for 10 minutes.

DETAILED DESCRIPTION:
Population 60 female during second stage of delivery

* Inclusion criteria : all parturients requiring pain relief will choose between systemic or epidural analgesia.
* Exclusion Criteria: all parturients with cardiac disease, neurological disease, endocrine disease, diabetes, hypertension or any parturients being treated with medications that might effect the cardiovascular autonomic system.
* Method: A 10 minute recording of a 3 lead ECG will be performed during the second stage of the delivery (3-7 CM opening).

the parturient will be lying on her left side for that period.

* 30 minutes after administration of either epidural or systemic Meperidine for pain relief, a second recording of maternal ECG will take place for 10 minutes.
* estimated duration of the procedure about one hour per woman.

ELIGIBILITY:
Inclusion Criteria: all parturients requiring pain relief will choose between systemic or epidural analgesia.

Exclusion Criteria: all parturients with cardiac disease, neurological disease, endocrine disease, diabetes, hypertension or any parturients being treated with medications that might effect the cardiovascular or autonomic system.

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Three lead ECG monitoring for 10 minutes will be performed 30 minutes after the administration.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Weissman, MD, Study Director — Rambam Health Care Campus; Olga Torchov, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam - health care campus, Haifa, Israel